CLINICAL TRIAL: NCT00859937
Title: Phase II Trial of Dasatinib (BMS 354825) for Recurrent or Metastatic c-KIT Expressing Adenoid Cystic Carcinoma and Non-adenoid Cystic Malignant Salivary Tumors
Brief Title: Dasatinib in Treating Patients With Recurrent or Metastatic Malignant Salivary Gland Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01165; NCI-2009-01165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000636685; UCCRC-16691B; 16691B (Other: University of Chicago Comprehensive Cancer Center); 8271 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Malignant Salivary Gland Neoplasm; Recurrent Salivary Gland Carcinoma; Salivary Gland Adenoid Cystic Carcinoma; Stage IV Major Salivary Gland Cancer AJCC v7
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Dasatinib

ARMS (1):
- Arm I (Experimental): Patients receive dasatinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well dasatinib works in treating patients with malignant salivary gland tumors that have come back after treatment or have spread to other parts of the body. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate (complete response plus partial response) of dasatinib in adenoid cystic carcinoma (ACC).

II. Determine the progression-free survival of dasatinib in ACC.

SECONDARY OBJECTIVES:

I. Determine the duration of response. II. Determine the stable disease rate and duration of stable disease. III. Determine progression-free survival. IV. Determine the median survival. V. Determine the overall survival. VI. Determine the safety and tolerability.

TERTIARY OBJECTIVES:

I. To examine biomarkers that relate to SRC proto-oncogene, non-receptor tyrosine kinase (Src) signal transduction and to correlate these biomarkers with clinical response to dasatinib in ACC and non-ACC malignant salivary gland tumors (MSGT).

II. Determine if activating mutations in platelet-derived growth factor alpha polypeptide (PDGFA) and KIT are associated with response in ACC.

OUTLINE:

Patients receive dasatinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant salivary gland tumor (MSGT), including one of the following histologic subtypes:

  * Adenoid cystic carcinoma (ACC) with c v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (Kit) overexpression or non-ACC MSGT that is not amenable to potentially curable surgery or radiation

    * c-KIT overexpression in ACC patients is defined as cluster of differentiation (CD) 117 staining by immunohistochemistry (IHC) in 25% of tumor cells
    * No stipulation for c-KIT overexpression is not required for non-ACC MSGT patients
* Patients must have radiographically measurable disease; radiographically measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients must have evidence of disease progression (objective growth of existing tumors) within 4 months of study entry
* No known brain metastases, unless patient meets both of the following criteria:

  * Neurologic status stable for >= 8 weeks after completion of definitive local therapy (surgery or radiotherapy)
  * No neurologic dysfunction that would confound study results
* Life expectancy greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 OR Karnofsky performance status (PS) >= 60%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Serum calcium =< 12.0 mg/dL
* Total serum bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; all women of childbearing potential must have a negative pregnancy test prior to receiving dasatinib; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; at least 4 weeks must have elapsed since any major surgery
* Patients may not be receiving any other investigational agents
* No prior treatment with any other targeted agents that inhibit vascular endothelial growth factor receptor (VEGFR), Breakpoint cluster region (BCR) ABL proto-oncogene 1, non-receptor tyrosine kinase (ABL), c-Src, c-KIT, platelet-derived growth factor (PDGF) beta receptor, or ephrin type-A receptor 2 (EPHA2) (e.g., imatinib mesylate)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib
* Patients with corrected QT interval (QTc) prolongation (defined as a QTc interval equal to or greater than 500 msec), serious ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia greater than or equal to 3 beats in a row) or other significant echocardiogram (ECG) abnormalities are excluded
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication, requirement for intravenous [IV] alimentation, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscesses within the past 28 days
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within the past 12 months
  * History of myocardial infraction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 6 months
  * History of pulmonary embolism within the past 12 months
  * Ejection fraction less than institutional normal by echocardiograph (only required for patients with a known history of congestive heart failure, low ejection fraction, or clinical symptoms/findings consistent with congestive heart failure)
* Patients taking medications that are potent inducers or inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) liver enzyme will be determined following a review of their case by the Principal Investigator; every effort should be made to switch patients taking such agents or substances to other medications
* Patients with known brain metastases should be excluded; patients with brain metastases with stable neurologic status following local therapy (surgery or radiation) for at least 8 weeks from definitive therapy and without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events are eligible for participation; patients cannot be receiving enzyme inducing anti-convulsants including carbamazepine, phenobarbital, and phenytoin
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with dasatinib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have an active pleural or pericardial effusion of any grade
* Diagnosis of any second malignancy within the last 5 years; basal cell carcinoma, squamous cell skin cancer, stage I carcinoma fully treated, or in situ carcinoma that have been adequately treated with no evidence of recurrent disease for 12 months will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03-16 (Actual); Primary Completion 2013-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Wong, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (34):
- United States (31):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM-Hotel Dieu de Montreal, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Adenoid Cystic Carcinoma: Patients with Adenoid cystic carcinoma of malignant salivary gland tumors receive oral dasatinib (70mg) twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Non Adenoid Cystic Carcinoma: Patients with non Adenoid cystic carcinoma of malignant salivary gland tumors receive oral dasatinib (70mg) twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Started | 41 | 14
Completed | 40 | 14
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma | Total
Number analyzed (Participants) | 40 | 14 | 54
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 82] | 56 [20 to 71] | 56 [20 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 4 | 26
  Male | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate is percentage of the best overall response which recoded from the start of the treatment until diseases progression/recurrence. Response criteria are defined using the international criteria proposed by the Response Evaluation Criteria In Solid Tumors (RECIST) Committee: Complete Response, Disappearance of all target lesions; Partial Response, >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease, neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: Up to 2 months
Population: There are two subtype cohorts, adenoid cystic carcinoma and non adenoid cystic carcinoma of malignant salivary gland tumors, with the same treatment. The two groups were analyzed separately and therefore no comparisons are made between the two groups.
Measure: Number; unit: participants
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Number analyzed (Participants) | 40 | 14
participants
  Complete response | 0 | 0
  Partial response | 1 | 0
  Stable disease | 20 | 7
  Progressive disease | 12 | 4
  Other | 7 | 3

2. Primary Outcome: Progression-free Survival
Description: Progression-free survival from start of treatment to the time of disease progression or death from any cause was estimated using the Kaplan-Meier method.
Time Frame: up to 5 years
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Number analyzed (Participants) | 40 | 14
months | 4.8 [1.9 to 5.5] | 2.7 [1.8 to 5.5]

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier curves will be generated and 90% confidence intervals will be derived.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Number analyzed (Participants) | 40 | 14
months | 14.5 [8.8 to 31.7] | 4.8 [2.2 to 8.0]

4. Secondary Outcome: Changes in Laboratory Correlates
Description: Changes in laboratory correlates pre-post therapy will be analyzed using paired t-tests. The association between RET gene rearrangements/mutations and tumor response, as well as the association between germ-line polymorp response, will be analyzed using Fisher's exact test. The correlative and genetic data will also be entered as cova only due to the small sample size) in a Cox regression model of progression-free survival.
Time Frame: Baseline and 4 weeks
Population: Biomarkers not done due to insufficient clinical responses thus making the biomarker analysis scientifically untenable.
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All serious adverse events were reported. Other adverse events occurring in ≥5% of the study subjects were reported.
Arm/Group | Adenoid Cystic Carcinoma | Non Adenoid Cystic Carcinoma
Serious Adverse Events (participants affected / at risk) | 12/40 | 8/14
Other Adverse Events (participants affected / at risk) | 39/40 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adenoid Cystic Carcinoma (N=40) | Non Adenoid Cystic Carcinoma (N=14)
Alanine aminotransferase increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections and infestations (Infections and infestations) | 1 | 0
Loss of vision (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adenoid Cystic Carcinoma (N=40) | Non Adenoid Cystic Carcinoma (N=14)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 10 | 4
Alkaline phosphatase increased (Investigations) | 7 | 0
Allergic reaction (Immune system disorders) | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 5
Anorexia (Metabolism and nutrition disorders) | 10 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Aspartate aminotransferase increased (Investigations) | 9 | 5
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Chills (General disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 11 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Creatinine increased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 13 | 6
Dizziness (Nervous system disorders) | 1 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Ear pain (Ear and labyrinth disorders) | 2 | 0
Edema face (General disorders) | 5 | 0
Edema limbs (General disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Eructation (Gastrointestinal disorders) | 0 | 1
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 24 | 9
Fever (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 16 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot flashes (Vascular disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2
INR increased (Investigations) | 0 | 1
Infections and infestations (Infections and infestations) | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 1
Libido decreased (Psychiatric disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 16 | 8
Neutrophil count decreased (Investigations) | 4 | 0
Nipple sensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 5 | 1
Oral pain (Gastrointestinal disorders) | 3 | 0
Pain (General disorders) | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Platelet count decreased (Investigations) | 7 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4
Weight loss (Investigations) | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
White blood cell decreased (Investigations) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less